CLINICAL TRIAL: NCT02903888
Title: A Cross-sectional, Observational Multicenter Study to Assess the Reasons for Choosing the 3-year Hormonal IUD and Level of IUDs Knowledge Among Women Aged 18 to 29 Years
Acronym: ANALIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18883
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Intrauterine Devices, Medicated
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BAY86-5028: Women aged 18 to 29 years that use Jaydess for contraception
  Interventions: Drug: Levonorgestrel (Jaydess, Skyla, BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel (Jaydess, Skyla, BAY86-5028) — Intrauterine delivery system Jaydess (13.5 mg levonorgestrel)

SUMMARY:
A cross-sectional, observational multicenter study to assess the reasons for choosing the 3-year hormonal IUD and level of IUDs knowledge among women aged 18 to 29 years. The study will be conducted in standard clinical practice conditions at public and private gynecology clinics and during a single study visit.

Approximately 1,000 women aged 18 to 29 years who have freely chosen the 3 year hormonal IUD as their contraceptive method will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 29 years.
* Women who decided to initiate treatment with a 3-year hormonal IUD for contraception after being adequately counseled and informed of all contraceptive options by their physician during a routine clinical visit, prior to the study visit (insertion visit).
* Women capable of reading and writing.
* Women who signed informed consent.

Exclusion Criteria:

* Women currently participating in an interventional clinical trial.
* Prescription of the 3-year hormonal IUD for non-contraceptive medical reasons.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of women aged 18-29 years, who have freely chosen Jaydess for contraception after being adequately counseled and informed of all contraceptive options by their physician at a previous visit to the study visit in a routine clinical practice setting
Sampling Method: Non-Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Reason for choosing Jaydess as intrauterine device (IUD) | day 1
  The participants select the reason out of a given list of 15 possible reasons
Reason for switching to Jaydess if used another type of intrauterine device before | day 1
  The participants select the reason out of a given list of 10 possible reasons
Knowledge of Jaydess or other IUDs prior to the visit | day 1
  The participants select the reason out of a given list of 3 possible reasons
Is the first intrauterine device prescribed? | day 1
  Possible reasons: Yes or No
Person who encouraged the use of jaydess? | day 1
  The participants select the answer out of a given list of 5 possible people

SECONDARY OUTCOMES:
Reason for not using Jaydess or other intrauterine delivery system (IUD) before | day 1
  The participants select the reason out of a given list of 12 possible reasons
Uterine length as measured by ultrasonography | day 1
Presence of dysmenorrhea (Y/N) | day 1
Current contraception method | day 1
  The participants select out of a given list of 20 options
Date of birth | day 1
Marital status | day 1
Place of birth | day 1
Place of residence | day 1
Educational level | day 1
Employment | day 1
Income level | day 1
Do you have children? (Y/N) | day 1
Number of children | day 1
Has she had some birth vaginally? (Y/N) | day 1
Date of last birth | day 1
Do you plan to have (more) children? (Yes/No/Unknown) | day 1
When she plans to have (more) children | day 1
Frequency of menstrual bleeding | day 1
Regularity of menstrual bleeding | day 1
Quantity of menstrual bleeding | day 1
Duration of menstrual bleeding | day 1
Absence of menstrual bleeding | day 1
Questionnaire concerning the physicians' characteristics | day 1
  The questionnaire consists of 7 questions

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Spain